CLINICAL TRIAL: NCT00283803
Title: Evaluation of the Effect of Exisulind on the Duration of the "Off-Treatment" Interval on Patients With Biochemical Relapse of Prostate Cancer Who Are Treated With Intermittent Androgen Suppression (ADT)
Brief Title: Exisulind and Intermittent Androgen Suppression (ADT) in Biochemical Relapsed Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Celestia Higano, Professor, Medicine, Division of Oncology & Urology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 44830; EX1006 (Other: OSI Pharmaceuticals)
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sulindac sulfone; Gonadotropin-Releasing Hormone; Leuprolide; Goserelin; Androgen Antagonists; Flutamide; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IAS and Exisulind (Experimental): Patients will receive intermittent dosing of hormone therapy with commercially supplied luteinizing hormone-releasing hormone (LHRH) agonist and anti-androgen to be chosen by physician per standard of care. Exisulind will be started 3 months prior to the end of the second cycle of hormone therapy. Patients will continue treatment with Exisulind beyond the completion of the second cycle of hormone therapy until they meet criteria for discontinuation.
  Interventions: Drug: Exisulind; Drug: luteinizing hormone-releasing hormone (LHRH) agonist; Drug: Antiandrogen

INTERVENTIONS:
Drug: Exisulind — Oral antineoplastic agent that induces apoptosis in cancerous cells.
  Other Names: Aptosyn
Drug: luteinizing hormone-releasing hormone (LHRH) agonist — Hormonal therapy to suppress testosterone as a standard treatment for Prostate Cancer.
  Other Names: Lupron; Zoladex
Drug: Antiandrogen — Hormonal therapy used as lead in treatment with luteinizing hormone-releasing hormone (LHRH) agonist to prevent the initial rise in testosterone (testosterone flare) seen during the first dose of LHRH agonists.
  Other Names: Eulexin; Casodex

SUMMARY:
The purpose of this research study is to determine if an investigational drug called Exisulind will extend the "off-treatment" period of patients receiving Intermittent Androgen Suppression (ADT).

There is evidence suggesting that alternating between periods of treatment and no treatment with androgen suppressants may delay the time to develop androgen-insensitive progression and improve overall quality of life. During intermittent androgen suppression (IAS) treatments, men receive a luteinizing hormone-releasing hormone (LHRH) agonist and antiandrogen for a fixed period of time (approximately 9 months) and then enter an off-treatment period, whose length will vary, depending on the rate of rise in the patient's Prostate-Specific Antigen (PSA). Once the PSA reaches an established threshold (1 ng/mL in men who have had a prostatectomy or 4 ng/ml in men with an intact prostate), androgen suppression will be re-initiated for another 9 months. These cycles of on-treatment/off-treatment will be repeated until patient no longer responds to the androgen suppression and it is clear that their cancer is progressing. It has been observed that off-treatment periods tend to become shorter with each successive cycle of androgen suppression, presumably due to the emergence of androgen-independent clones. This study proposes to look at exisulind, a pro-apoptotic drug, which may extend the off-treatment period in patients receiving IAS.

DETAILED DESCRIPTION:
A study doctor will meet with you and ask you about your medical history, examine you, and explain the study. We will draw some blood for tests (about 4-6 tablespoons), including Prostate-Specific Antigen (PSA). If not already obtained, you will have a bone scan and a computed tomography scan (CT scan) to establish a baseline.

You will be receiving hormone suppression treatment with monthly injections of a luteinizing hormone-releasing hormone (LHRH) analog such as Lupron or Zoladex and an antiandrogen such as Eulexin or Casodex as part of your standard care for prostate cancer. About 3 months before your next "off-treatment" period, you will start 1 Exisulind pill 250 mg (2 x 125mg capsules) by mouth twice a day. It is necessary for you to start the Exisulind treatment 3 months prior to your next "off-treatment" period so that the medication can build up in your system enough to be effective.

Per our standard follow-up procedures, we will ask you to have blood draws every 2 weeks for up to 12 weeks after starting Exisulind to check liver function. Thereafter you will be asked to have monthly blood draws, and return to the clinic every 3 months for a physical examination, to determine how well you are tolerating the study medication, how your cancer is responding to the treatment, and to give you more study medication. You will continue taking Exisulind during your "off-treatment" period until your PSA reaches a threshold level. PSA threshold is defined by your primary treatment. If you have had your prostate removed, the threshold is 1.0 ng/dL. If you have an intact prostate, your threshold is 4 ng/dL. Once your PSA reaches this level, you will restart your hormone suppression treatment as directed by your doctor.

ELIGIBILITY:
Inclusion Criteria:

* A willingness and ability to sign an informed consent document;

  * 21 years or of legal age;
* Histologically or cytologically documented prostate cancer.
* ECOG Performance status score of 0 or 1.
* Received at least one cycle of IAS with an LHRH agonist and anti-androgen
* Willingness to remain off chronic NSAIDs (with the exception of ibuprofen or naproxen), including COX 2 inhibitors and salicylates (e.g., aspirin, mesalamine, azodisalicylate, salsalate, sulfasalazine) for duration of the study. Patients on low dose aspirin for cardiovascular prevention may be included in the study.
* Have not taken sulindac (Clinoril™) on regular basis for any indication for one week prior to enrollment and willing to remain off of sulindac for the duration of the study.
* Patients with prior radiation must be 2 weeks from their last radiation-treatment and have recovered from all associated toxicity.

Exclusion Criteria:

* Known hypersensitivity to sulindac (Clinoril™)
* ECOG Performance status score > 1;
* Patients previously on SWOG 9346 or 9921 trials, or any other trials using IAS for which adding exisulind may be confounding.
* Patients may not have any evidence of hormone-refractory prostate cancer, i.e. 2 consecutive rises in PSA on LHRH agonist and anti-androgen
* Active peptic ulcer disease;
* Use of an investigational medication or device within one month of initiating study therapy;
* Elevations of serum creatinine to above the upper limit of normal;
* Platelet count < 100,000/L; hgb < 9.0 g/dL; absolute neutrophil count < 1500/mm3
* Known hepatic, biliary tract, renal or hematologic dysfunction which in the opinion of the Investigator or Sponsor are clinically significant or would obscure laboratory analyses or are associated with lab abnormalities;
* Any condition or any medication that may interfere with the conduct of the study.
* Bilirubin > ULN. Patients with elevated indirect bilirubin due to Gilbert's Syndrome will be eligible.
* AST or ALT >2.5 X ULN

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-03-12 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celestia Higano, MD, Principal Investigator — University of Washington
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrolled 32 subjects who had developed biochemical progression of prostate cancer, shown by the rising prostate specific antigen level (PSA) after curative therapy (either a radical prostatectomy or external beam irradiation). Trial was open to enrollment 2002 through 2004.
Pre-assignment Details: Approximately 40 patients were considered. A total of 32 were accrued between 12Mar2002 and 29Oct2004. Patients not enrolled either failed to meet eligibility criteria or withdrew consent prior to treatment. 19 patients completed study and were evaluable for study endpoints.
Groups:
- Exisulind: Patients will receive intermittent dosing of hormone therapy with commercially supplied LHRH agonist and antiandrogen to be chosen by physician per standard of care. Exisulind will be started 3 months prior to the end of the second cycle of hormone therapy. Patients will continue treatment with Exisulind beyond the completion of the second cycle of hormone therapy until they meet criteria for discontinuation.
  Exisulind: Exisulind 125 mg
Period: Overall Study
Arm/Group | Exisulind
Started | 32
Completed | 19
Not Completed | 13
Not completed — Physician Decision | 9
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- IAS and Exisulind: Patients will receive intermittent dosing of hormone therapy with commercially supplied LHRH agonist and antiandrogen to be chosen by physician per standard of care. Exisulind will be started 3 months prior to the end of the second cycle of hormone therapy. Patients will continue treatment with Exisulind beyond the completion of the second cycle of hormone therapy until they meet criteria for discontinuation.
Arm/Group | IAS and Exisulind
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Duration of the First "Off-treatment" Cycle in Patients Who Have Completed One Cycle of Intermittent Androgen Suppression With the Addition of Exisulind.
Description: Patients were monitored for the amount of time (number of weeks) that passed between the completion of a cycle of Intermittent Androgen Suppression with Exisulind and the need to re-initiate treatment with Intermittent Androgen Suppression. It was hoped that adding Exisulind to standard Androgen Suppression would extend the amount time before disease progression.
Time Frame: From date of first treatment until the date of first documented progression or study withdrawal, whichever came first, assessed up to 10 years.
Population: Of the 32 patients who enrolled, 19 were evaluable.
Measure: Mean (Full Range); unit: Weeks
Arm/Group | IAS and Exisulind
Number analyzed (Participants) | 19
Weeks | 39 [25 to 71]

2. Primary Outcome: Time to Hormone-refractory Diseases in Patients Treated With Intermittent Androgen Suppression and Exisulind
Description: Patients were monitored for continued hormonal sensitivity of their disease from the time of the first treatment with Intermittent Androgen Suppression and Exisulind and the time at which point they were considered hormone-refractory (castrate resistant). The development of hormone-refractory disease was one of the criteria for withdraw from study treatment. For this protocol, hormone-refractory was defined as 2 consecutive rising PSAs at least 2 weeks apart while on an LHRH agonist (with or without an anti-androgen).
Time Frame: as for outcome 1
Population: Out of 32 enrolled patients, 19 met criteria to be evaluable.
Measure: Median (Full Range); unit: Weeks
Arm/Group | IAS and Exisulind
Number analyzed (Participants) | 19
Weeks | 286 [15.6 to NA] — Maximum range of time to CRPC is N/A because some patients did not become Castrate Resistant prior to end of study.

3. Primary Outcome: Number of Participants With Dose Hold, Dose Reduction, or Treatment Withdrawal for Toxicity.
Description: Patients were monitored for toxicity related treatment modifications from the start of Exisulind through the time that there were withdrawn from study.
Time Frame: From date of first treatment until study withdrawal, assessed up to 10 years.
Population: Of 32 enrolled patients, 19 met criteria to be evaluable for study.
Measure: Count of Participants; unit: Participants
Arm/Group | IAS and Exisulind
Number analyzed (Participants) | 19
Participants
  Dose Hold for Toxicity | 6
  Dose Reduction for Toxicity | 9
  Treatment Withdrawn for Toxicity | 7

ADVERSE EVENTS:
Time Frame: Adverse Events collected for each patient from time of starting Exisulind through time of study withdraw, assessed up to 10 years.
Description: The term "adverse event" could include any of the following events that arise or increase in severity and/or frequency during the course of the study:
  * signs or symptoms
  * clinically significant laboratory abnormality
  * abnormality detected during physical exam
  These data will be recorded regardless of whether they are thought to be associated with the study or the drug under investigation.
Arm/Group | Exisulind
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 21/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exisulind (N=32)
Gallstone with cholecystectomy (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) — One patient was hospitalized from loss of consciousness and was ultimately diagnosed with pneumonia. The patient was discharged after 1 day and it was determined that this event was not related to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exisulind (N=32)
Elevated LFTs (Investigations) | 10
Fatigue (General disorders) | 8
Nocturia (Renal and urinary disorders) | 7
Hot Flashes (General disorders) | 7
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 6
Congested Sinuses/Cold (Infections and infestations) | 6
Anemia (Investigations) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Hypertriglyceridemia/Hyperlipidemia (Investigations) | 5
Renal Insufficiency (Renal and urinary disorders) | 4
Pain/Soreness/Cramps - leg(s) (Musculoskeletal and connective tissue disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3
Weight loss (Metabolism and nutrition disorders) | 3
Hypertension (Cardiac disorders) | 3
Depression (Psychiatric disorders) | 3
Weight Gain (Metabolism and nutrition disorders) | 3
Decreased Libido (Reproductive system and breast disorders) | 3

LIMITATIONS AND CAVEATS:
Enrollment goal was 35 evaluable patients. Of the 40+ considered, 32 consented and enrolled. However 13 withdrew, leaving only 19 evaluable patients. Due to small sample size, results were primarily descriptive in nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No